CLINICAL TRIAL: NCT06034743
Title: A Randomised, Double-Blind, Placebo-Controlled, Parallel Group Study to Assess the Efficacy and Safety of Baxdrostat in Participants With Uncontrolled Hypertension on Two or More Medications Including Participants With Resistant Hypertension
Brief Title: A Study to Investigate the Efficacy and Safety of Baxdrostat in Participants With Uncontrolled Hypertension on Two or More Medications Including Participants With Resistant Hypertension
Acronym: BaxHTN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6970C00002; 2023-505499-32-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2023-09-06; First posted 2023-09-13 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Uncontrolled Hypertension; Resistant Hypertension
Keywords: Hypertension; Uncontrolled hypertension; Resistant hypertension; Blood pressure; Baxdrostat; CIN-107; Aldosterone; Aldosterone synthase
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 2 mg baxdrostat (Experimental): 2 mg baxdrostat administered orally, once daily (QD).
  Interventions: Drug: Baxdrostat
- 1 mg baxdrostat (Experimental): 1 mg baxdrostat administered orally, once daily (QD).
  Interventions: Drug: Baxdrostat
- Placebo (Placebo Comparator): Placebo administered orally, once daily (QD).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baxdrostat — Baxdrostat tablet administered orally, once daily (QD). Unit dose strengths:
  * 1 mg per tablet for 1 mg baxdrostat Arm;
  * 2 mg per tablet for 2 mg baxdrostat Arm.
  Other Names: CIN-107
  Arms: 1 mg baxdrostat; 2 mg baxdrostat
Drug: Placebo — Placebo tablet matching baxdrostat, administered orally, once daily (QD).
  Arms: Placebo

SUMMARY:
This is a Phase III, multicentre, randomised, double-blinded, placebo-controlled, parallel group study to evaluate the safety, tolerability and effect of 1 or 2 mg baxdrostat versus placebo, administered once daily (QD) orally, on the reduction of systolic blood pressure in approximately 720 participants aged ≥ 18 years with hypertension, despite a stable regimen of 2 antihypertensive agents at baseline, one of which is a diuretic (uncontrolled hypertension); or ≥ 3 antihypertensive agents at baseline, one of which is a diuretic (treatment-resistant hypertension).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants must be ≥ 18 years old
* Mean sitting systolic blood pressure on automated office blood pressure measurement ≥ 140 mmHg and < 170 mmHg at Screening
* Fulfil at least 1 of the following 2 criteria:

  1. uHTN subpopulation: have a stable regimen of 2 antihypertensive medications, from different therapeutic classes (at least one must be a diuretic), at maximum tolerated dose in the judgement of the Investigator
  2. rHTN subpopulation: have a stable regimen of ≥ 3 antihypertensive medications, from different therapeutic classes (at least one must be a diuretic), at maximum tolerated dose in the judgement of the Investigator
* Estimated glomerular filtration rate ≥ 45 mL/min/1.73m2 at Screening
* Serum potassium (K+) level ≥ 3.5 and < 5.0 mmol/L at Screening
* Randomisation Criterion:
* Sitting systolic blood pressure on attended automated office blood pressure measurement of ≥ 135 mmHg at the Baseline Visit

Exclusion Criteria:

* Mean sitting systolic blood pressure on attended automated office blood pressure measurement ≥ 170 mmHg
* Mean seated diastolic blood pressure on attended automated office blood pressure measurement ≥ 110 mmHg
* Serum sodium level < 135 mmol/L at Screening
* Has the following known secondary causes of hypertension: renal artery stenosis, uncontrolled or untreated hyperthyroidism, uncontrolled or untreated hypothyroidism, pheochromocytoma, Cushing's syndrome, aortic coarctation
* New York Heart Association functional heart failure class IV at Screening
* Persistent atrial fibrillation

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 796 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in seated systolic blood pressure for 2 mg baxdrostat | At Week 12
  To assess the effect of 2 mg baxdrostat versus placebo on seated systolic blood pressure at Week 12
Change from baseline in seated systolic blood pressure for 1 mg baxdrostat | At Week 12
  To assess the effect of 1 mg baxdrostat versus placebo on seated systolic blood pressure at Week 12

SECONDARY OUTCOMES:
Change from randomised withdrawal baseline (Week 24) in seated systolic blood pressure (SBP) for 2 mg baxdrostat | At Week 32
  To assess the effect of 2 mg baxdrostat vs placebo on seated systolic blood pressure (SBP) at 8 weeks after randomised withdrawal
Change from baseline in seated SBP for 2 mg baxdrostat | At Week 12
  To assess the effect of 2 mg baxdrostat vs placebo on seated SBP at Week 12 in the resistant hypertension (rHTN) subpopulation
Change from baseline in seated diastolic blood pressure (DBP) for 2 mg baxdrostat | At Week 12
  To assess the effect of 2 mg baxdrostat vs placebo on seated diastolic blood pressure (DBP) at Week 12
Achieving seated SBP < 130 mmHg for 2 mg baxdrostat | At Week 12
  To assess the effect of 2 mg baxdrostat vs placebo on achieving seated SBP < 130 mmHg at Week 12
Change from baseline in seated SBP for 1 mg baxdrostat | At Week 12
  To assess the effect of 1 mg baxdrostat vs placebo on seated SBP at Week 12 in the rHTN subpopulation
Change from baseline in seated DBP for 1 mg baxdrostat | At Week 12
  To assess the effect of 1 mg baxdrostat vs placebo on seated DBP at Week 12
Achieving seated SBP < 130 mmHg for 1 mg baxdrostat | At Week 12
  To assess the effect of 1 mg baxdrostat vs placebo on achieving seated SBP < 130 mmHg at Week 12

OTHER OUTCOMES:
Number of participants with adverse events (AEs) | Up to Week 54
  To assess the safety and tolerability of baxdrostat versus placebo. Occurrence of adverse events (AE), including serious adverse events (SAEs), adverse events leading to treatment discontinuation (DAE) and adverse events of special interest (AESI).

CONTACTS AND LOCATIONS:
Locations (225):
- United States (41):
  - Research Site, Saraland, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Sun City West, Arizona
  - Research Site, Surprise, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Fresno, California
  - Research Site, Lincoln, California
  - Research Site, Orange, California
  - Research Site, Rancho Cucamonga, California
  - Research Site, Stanford, California
  - Research Site, New Haven, Connecticut
  - Research Site, Clearwater, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Port Orange, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Decatur, Georgia
  - Research Site, Springfield, Illinois
  - Research Site, Munster, Indiana
  - Research Site, Lexington, Kentucky
  - Research Site, Detroit, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, Olive Branch, Mississippi
  - Research Site, Kansas City, Missouri
  - Research Site, Rosedale, New York
  - Research Site, The Bronx, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Toledo, Ohio
  - Research Site, Grants Pass, Oregon
  - Research Site, Bethlehem, Pennsylvania
  - Research Site, Langhorne, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Memphis, Tennessee
  - Research Site, Brownsville, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Houston, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Manassas, Virginia
  - Research Site, Suffolk, Virginia
  - Research Site, Madison, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Argentina (9):
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Córdoba
  - Research Site, Mar del Plata
  - Research Site, Mendoza
  - Research Site, Rosario
  - Research Site, San Miguel de Tucumán
  - Research Site, San Nicolás
  - Research Site, San Vicente
- Australia (9):
  - Research Site, Clayton
  - Research Site, Darlinghurst
  - Research Site, Epping
  - Research Site, Geelong
  - Research Site, Liverpool
  - Research Site, New Lambton Heights
  - Research Site, Perth
  - Research Site, Wollongong
  - Research Site, Woolloongabba
- Austria (3):
  - Research Site, Braunau am Inn
  - Research Site, Sankt Pölten
  - Research Site, Vienna
- Belgium (3):
  - Research Site, Ghent
  - Research Site, Liège
  - Research Site, Mons
- Bulgaria (2):
  - Research Site, Pleven
  - Research Site, Sofia
- Canada (11):
  - Research Site, Edmonton, Alberta
  - Research Site, North Vancouver, British Columbia
  - Research Site, Cambridge, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Saint-Jean-sur-Richelieu, Quebec
- Czechia (7):
  - Research Site, Benešov
  - Research Site, Brandýs nad Labem
  - Research Site, Broumov
  - Research Site, Louny
  - Research Site, Ostrava
  - Research Site, Příbram
  - Research Site, Uherské Hradiště
- Denmark (3):
  - Research Site, Aarhus
  - Research Site, Herning
  - Research Site, Holbæk
- France (7):
  - Research Site, Bobigny
  - Research Site, Bordeaux
  - Research Site, Paris
  - Research Site, Saint-Priest-en-Jarez
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tours
- Germany (15):
  - Research Site, Bad Homburg
  - Research Site, Bad Oeynhausen
  - Research Site, Berlin
  - Research Site, Dortmund
  - Research Site, Düsseldorf
  - Research Site, Elsterwerda
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Hanover
  - Research Site, Homburg
  - Research Site, Kaiserslautern
  - Research Site, Leipzig
  - Research Site, Mannheim
  - Research Site, Wermsdorf
- Hungary (6):
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Kalocsa
  - Research Site, Kaposvár
  - Research Site, Nyíregyháza
  - Research Site, Pécs
- India (7):
  - Research Site, Delhi
  - Research Site, Guntur
  - Research Site, Kanpur
  - Research Site, Kolkata
  - Research Site, Mysuru
  - Research Site, New Delhi
  - Research Site, Surat
- Israel (5):
  - Research Site, Ashdod
  - Research Site, Haifa
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Rehovot
- Italy (8):
  - Research Site, Acquaviva delle Fonti
  - Research Site, Bologna
  - Research Site, Brescia
  - Research Site, Milan
  - Research Site, Pisa
  - Research Site, Roma
  - Research Site, Torino
  - Research Site, Udine
- Japan (11):
  - Research Site, Adachi-ku
  - Research Site, Chūōku
  - Research Site, Kanazawa
  - Research Site, Koga-shi
  - Research Site, Kyoto
  - Research Site, Nagasaki
  - Research Site, Okayama
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Tsuchiura-shi
  - Research Site, Yufu-shi
- Malaysia (7):
  - Research Site, Kajang
  - Research Site, Kota Bharu
  - Research Site, Kuching
  - Research Site, Malacca
  - Research Site, Muar town
  - Research Site, Sarawak Miri
  - Research Site, Seri Manjung
- Netherlands (3):
  - Research Site, Hoogeveen
  - Research Site, Nijmegen
  - Research Site, Utrecht
- Poland (9):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Chrzanów
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Warsaw
- Slovakia (6):
  - Research Site, Brezno
  - Research Site, Košice
  - Research Site, Moldava nad Bodvou
  - Research Site, Prešov
  - Research Site, Rimavská Sobota
  - Research Site, Svidník
- South Africa (7):
  - Research Site, Cape Town
  - Research Site, Centurion
  - Research Site, Claremont
  - Research Site, Durban
  - Research Site, Kwadwesi
  - Research Site, Somerset West
  - Research Site, Worcester
- South Korea (5):
  - Research Site, Bucheon-si
  - Research Site, Busan
  - Research Site, Daejeon
  - Research Site, Incheon
  - Research Site, Seoul
- Spain (7):
  - Research Site, Barcelona
  - Research Site, Ferrol
  - Research Site, Granada
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Seville
  - Research Site, Terrassa (Barcelona)
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Uppsala
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Yung Kang City
- Thailand (5):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Pathum Thani
- Turkey (Türkiye) (8):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Bursa
  - Research Site, Dinar
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kütahya
  - Research Site, Odunpazari
- United Kingdom (11):
  - Research Site, Bollington
  - Research Site, Bristol
  - Research Site, Chesterfield
  - Research Site, Dundee
  - Research Site, Glasgow
  - Research Site, Harrow
  - Research Site, Hownslow
  - Research Site, London
  - Research Site, Prescot
  - Research Site, Weston-super-Mare
  - Research Site, Yate
- Vietnam (4):
  - Research Site, Da Nang
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Flack JM, Azizi M, Brown JM, Dwyer JP, Fronczek J, Jones ESW, Olsson DS, Perl S, Shibata H, Wang JG, Wilderang U, Wittes J, Williams B; BaxHTN Investigators. Efficacy and Safety of Baxdrostat in Uncontrolled and Resistant Hypertension. N Engl J Med. 2025 Oct 9;393(14):1363-1374. doi: 10.1056/NEJMoa2507109. Epub 2025 Aug 30. PMID 40888730